CLINICAL TRIAL: NCT07259798
Title: Comparison Between En-Bloc Transurethral Resection Versus Conventional Transurethral Resection of Urinary Bladder Tumors From 2 to 6 cm in Size, Histopathological Findings.
Brief Title: Histopathological Findings in En-Bloc vs Conventional Transurethral Resection of Bladder Tumors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Younan Ramsis, Lecturer of Urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FMASU MS429/2024
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Urinary Bladder Cancer
Keywords: TURBT; en bloc TURBT; TCC of the bladder; Histopathological findings
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Underwent En bloc Bipolar TURBT (Experimental)
  Interventions: Procedure: En bloc TURBT using a bipolar Karl-Storz resectoscope system fitted with a specialized "flat" resection loop
- Group B: Bipolar piecemeal TURBT (Active Comparator)
  Interventions: Procedure: Bipolar piecemeal TURBT using the same bipolar Karl-Storz resectoscopic platform

INTERVENTIONS:
Procedure: En bloc TURBT using a bipolar Karl-Storz resectoscope system fitted with a specialized "flat" resection loop — A specialized "flat" resection loop (Karl-Storz En-Bloc Electrode, stainless steel, approximately 24 mm diameter). This loop features a broad, planar configuration with a smooth leading edge designed to dissect beneath the tumor base in a single piece while maintaining an intact specimen-muscle interface and minimizing fragmentation.
  Arms: Group A: Underwent En bloc Bipolar TURBT
Procedure: Bipolar piecemeal TURBT using the same bipolar Karl-Storz resectoscopic platform — The resections were performed with a standard U-shaped cutting loop electrode (Karl-Storz, stainless steel, 24 mm diameter) mounted on a bipolar working element compatible with a 26-Fr continuous-flow resectoscope sheath and a 30-degree Hopkins® rod-lens telescope. The U-shaped loop, characterized by its semi elliptical contour and dual active cutting arms, facilitates sequential layer-by-layer resection of the tumor in multiple fragments, permitting simultaneous coagulation of bleeding vessels.
  Arms: Group B: Bipolar piecemeal TURBT

SUMMARY:
This study is designed to determine whether en-bloc TURBT provides superior histopathological quality and clinical outcomes compared to conventional TURBT in medium-sized bladder tumors.

DETAILED DESCRIPTION:
This study is a prospective randomized clinical trial conducted at Ain Shams University to compare en-bloc transurethral resection (ERBT) with conventional transurethral resection (TURBT) for urinary bladder tumors sized 2-6 cm. The primary endpoint is the presence of detrusor muscle in histopathological specimens, while secondary outcomes include bladder perforation, residual disease at second TURBT, margin status, operation time, obturator reflex, and conversion rates. By focusing on specimen integrity and surgical efficacy, the study aims to determine whether en-bloc TURBT provides superior diagnostic accuracy and clinical outcomes compared to the conventional approach.

ELIGIBILITY:
Inclusion Criteria:

* Tumor diameter of 2-6 cm
* Patients fit for spinal or general anesthesia

Exclusion Criteria:

* recurrent bladder tumours.
* concomitant urothelial cancer of the upper urinary tract
* metastatic bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
the presence of detrusor muscle in histopathologic specimens | 10 days post TURBT
  This assessment aims to compare the histopathological outcomes between the tumors obtained from the en bloc bipolar resection versus the conventional method bipolar Trans-Urethral Resection of Bladder Tumor techniques

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed K Ahmed, Assisstant Professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yang H, Lin J, Gao P, He Z, Kuang X, Li X, Fu H, Du D. Is the En Bloc Transurethral Resection More Effective than Conventional Transurethral Resection for Non-Muscle-Invasive Bladder Cancer? A Systematic Review and Meta-Analysis. Urol Int. 2020;104(5-6):402-409. doi: 10.1159/000503734. Epub 2020 Jan 7. PMID 31910427
- [Result] Sun S, Wang H, Zhang X, Chen G. Transurethral Resection of Bladder Tumor: Novel Techniques in a New Era. Bladder (San Franc). 2023 Nov 9;10:e21200009. doi: 10.14440/bladder.2023.865. eCollection 2023. PMID 38022709